CLINICAL TRIAL: NCT05390645
Title: An Open-label, Multi-center, Phase I/II Study of MFA-370 in Patients with Metastatic Urothelial Cancer
Brief Title: A Study of MFA-370 in Patients with Metastatic Urothelial Cancer
Acronym: MANHATTAN
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor company was liquidated.
Sponsor: Ectin Research AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ECT-001; 2021-000068-30 (EudraCT Number)
Record Dates: First submitted 2022-03-09; First posted 2022-05-25 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Urothelial Cancer
Keywords: Metastatic Urothelial Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MFA-370 (Experimental): MFA-370 once daily for up to 8 x 21 days.
  Interventions: Drug: MFA-370

INTERVENTIONS:
Drug: MFA-370 — MFA-370 is a treatment with a combination of two approved pharmaceuticals

SUMMARY:
This is a multi-center study of MFA-370 in patients with metastatic urothelial cancer. The objective of the study is to assess the safety and efficacy of MFA-370, i.e.a combination of two approved pharmaceuticals today used within other indications. The combination was developed after the finding that a multidiseased man with e.g. muscle-invasive bladder cancer also was treated for his recent parasitic infection resulted in that the parasitic infection together with the cancer got a complete remission. After extensive experimental complementing studies a combination treatment called MFA-370 was developed supporting the rationale for this treatment.

This is the first clinical trial where the combination product MFA-370 is evaluated as anti-cancer treatment. Up to 50 patients will participate.

MFA-370 is taken orally once daily for up to 24 weeks. If the treatment is of clinical benefit for the patient, as assessed by the investigator, the treatment period can be prolonged to up to 2 years.

The patients will be monitored for safety, tolerability, pharmacokinetics, tumor response by RECIST (Response Evaluation Criteria in Solid Tumors) 1.1 and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form before any screening procedures
2. ≥ 18 years of age on the day of giving informed consent
3. Confirmed current metastatic urothelial carcinoma of the bladder, including the urethra and upper urinary tract. The patient needs to have progressive disease and/or symptomatic metastatic disease that is unresponsive to standard therapy. The patient must have received all available approved therapies before being eligible for the study unless contraindications or intolerance exist for one or several of them
4. At least one lesion of measurable disease as defined by RECIST1.1 criteria based on CT or MRI scan within 2 weeks before start at Day -7
5. World Health Organization (WHO) performance status 0-2
6. Life expectancy ≥12 weeks
7. Patients with reproductive potential will need to use accepted and highly effective means of contraception from study entry until at least 6 weeks for females (women of childbearing potential) and 3 months for males after study drug discontinuation

Main Exclusion Criteria:

1. Known CNS metastatic lesions, or evidence of impaired blood-brain barrier as assessed by the investigator
2. Have signs or symptoms of active COVID-19 infection or a positive COVID-19 Polymerase Chain Reaction (PCR) test during the screening period
3. Impaired renal function by estimated Glomerular Filtration Rate (eGFR) <30 ml/min as per local assessment
4. Laboratory values (hematology and biochemistry) within specified ranges to show appropriate organ function
5. Clinically significant cardiac disease,
6. Untreated or uncontrolled hypertension
7. An underlying medical condition that precludes the ability to take oral medication daily
8. Prohibited concomitant therapy
9. The patient has had biologic, hormonal, anti-neoplastic chemotherapy, or radiation therapy other than palliative treatment within 4 weeks prior to screening except for medications with half-lives <5.5 days
10. Hypersensitivity to the active ingredients or to any of the excipients listed in section 6.1 in respective Summary of Product Characteristics (SmPC)
11. Any bleeding disorder or condition where there is an increased risk of bleeding
12. A history of allergic reactions following intake of acetylsalicylic acid or NSAIDs
13. A history of gastrointestinal bleeding or perforation
14. Active or recurrent gastrointestinal ulcer
15. Major surgery within 14 days before enrolment. (Note: trans-urethral resection of bladder tumor is not considered major surgery)
16. For female patients of childbearing potential - pregnancy, as confirmed by a serum pregnancy test at screening, or breast-feeding
17. Any other severe, acute, or chronic medical condition that would interfere with the conduct of the study or interpretation of the study results as judged by the investigator
18. The patient has already participated in the study or been a screening failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | Up to 30 days safety follow up
  Safety of MFA-370 measured by incidence and severity of AEs and serious SAEs with a causal relationship to MFA-370
Incidence of dose interruptions, reductions, and treatment terminations due to AEs/SAEs | Up to 30 days safety follow up
  Tolerability of MFA-370 measured by incidence of dose interruptions, reductions, and treatment terminations due to AEs/SAEs
Overall Response Rate (ORR) | At 24 weeks
  Anti-tumor activity of MFA-370 measured by Overall Response Rate (ORR), assessed by the investigator based on the assessment of the Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) scans made by the responsible Radiologist at each site (scans assessed per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1)

SECONDARY OUTCOMES:
Overall Response Rate (ORR), Clinical Benefit Rate (CBR), Progression-Free Survival (PFS), Time to Progression (TTP), Best Overall Response (BOR) | Every six weeks up to 24 weeks
  Anti-tumor activity of MFA-370 measured by ORR, CBR, PFS, TTP, BOR based on CT/MRI-scans assessed by Radiologist per RECIST 1.1
Incidence and severity of AEs and SAEs | Up to 30 days after last dose
  Safety of MFA-370 measured by incidence and severity of AEs and SAEs with a causal relationship to MFA-370
Incidence of dose interruptions, reductions, and treatment terminations due to AEs/SAEs | Up to 30 days after last dose
  Tolerability of MFA-370 measured by incidence of dose interruptions, reductions, and treatment terminations due to AEs
Overall Survival | From the last dose until the date of death or up to 6 months after the last patient's end of treatment, whichever came first.
  Effect of MFA-370 on Overall Survival
Plasma concentration profiles | From start of treatment until 29th day of treatment
  To characterize the pharmacokinetic properties of MFA-370 with respect to time vs plasma concentration profiles
Peak Plasma Concentration (Cmax) | From start of treatment until 29th day of treatment
  To characterize the pharmacokinetic properties of MFA-370 with respect to Cmax in plasma
Time to reach peak plasma concentration (tmax) of MFA-370 in plasma | From start of treatment until 29th day of treatment
  To characterize the pharmacokinetic properties of MFA-370 with respect to tmax
Elimination half-life (t1/2) of MFA-370 in plasma | From start of treatment until 29th day of treatment
  To characterize the pharmacokinetic properties of MFA-370 with respect to t1/2

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden